CLINICAL TRIAL: NCT01862809
Title: The Effect of Smoking on Oral Microbiota
Brief Title: Cigarette Smoking and Oral Microbiota
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999913103; 13-C-N103
Record Dates: First submitted 2013-05-23; First posted 2013-05-24 (Estimated); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Microbiota; Lung Cancer; Oral Cancer
Keywords: Oral Microbiota; Cigarette Smoking; Tobacco- Related Cancer
MeSH Terms: conditions — Lung Neoplasms; Mouth Neoplasms; Cigarette Smoking

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other

GROUPS / COHORTS (2):
- cases: smokers
- controls: non-smokers

SUMMARY:
Background:

- Normal bacteria and other tiny organisms (the microbiota) live in the mouth and nose. They contribute to human health in many ways, including digesting food and balancing hormones. Testing samples from the mouth can show how microbiotas are related to health and disease. However, the microbiota in a person's mouth differs depending on the methods of collection and the part of the mouth that is tested. Understanding what can change the microbiota (including mouth sites, and what a person eats or smokes) will give more information on how to study oral microbiota and smoking-related cancers and other diseases.

Objectives:

* To see how smoking affects the microbiotas in mouth and nose.
* To determine which collection method for mouth specimens should be used for studying microbiota.

Eligibility:

* Individuals at least 18 years of age who have been using tobacco products regularly for at least 5 years.
* Individuals at least 18 years of age who have never smoked.

Design:

* Participants will be screened with a physical exam and medical history.
* Participants will have a dental exam. They will provide a saliva sample. The dentist will take swabs from the inside of the mouth, including the tongue, tonsils, gums, and teeth. The inside of the nose will also be swabbed.
* Participants will also fill out a questionnaire. It will ask about their history of smoking and consumption of alcohol, tea, and coffee. It will also ask about current medications, including antibiotics.

DETAILED DESCRIPTION:
The oral microbial community (the microbiota), is centrally related to nutrition, metabolism, immunity, inflammation, and endocrine balance. Cigarette smoking is associated with serious health outcomes including cancer, cardiovascular disease and chronic lung disease. However, little is known about the relationship between cigarette smoking, oral microbiota and tobacco-related health outcomes. Microbiotas in the different sites of the same oral cavity vary widely. Recent studies indicated that the difference in microbial profiles between buccal mucosa and gingival plaque is as distinct as the difference between tongue and stool. To date, knowledge about the effect of smoking on oral microbiotas is lacking. As an initial step toward understanding the role of the oral microbiota in smoking-related health outcomes, we propose a pilot study to evaluate the effects of cigarette smoking on the microbiotas in buccal rinse obtained from the oral cavity and across 8 different oral cavity sites/niches (saliva, swabs from tongue dorsum, hard palate, buccal mucosa, keratinized gingiva, palatine tonsils, supragingival plaque, subgingival plaque). We will seek to recruit up to 50 volunteers through the Eastman Dental General Dentistry Clinic, Rochester, NY, including 25 current smokers with > 5 years of smoking history and 25 never smokers as a comparison group. Age-group, gender, and race (Caucasian/African- American) will be matched for the two groups. In each subject, the buccal cell (mouthwash) collection will be collected according to the PLCO buccal cell collection protocol. In addition, collections across 8 different oral cavity sites will be done using a protocol developed for the Human Microbiome Project. These 9 collections will be used for high throughput sequencing of 16S rRNA microbial genes at the Institute of Genome Sciences, University of Maryland School of Medicine. The findings will provide information about the effect of smoking on microbial taxa composition and relative abundance at each collection site. This pilot study will demonstrate the effects of smoking on oral microbiotas across different oral cavity sites and will also demonstrate which oral collection site is most promising for the detailed study about cigarette smoking and oral microbiota. In addition, the data collected will provide a validation framework to use the PLCO buccal specimens for large-scale studies. The information about the validity of using PLCO buccal cell collection will be an invaluable asset for further large scale studies of the microbiota and cancer risk. We will also be able to investigate if there is any taxonomy or microbial diversity difference between heavy smokers and never-smokers. This pilot study will provide essential information about collection, design and analyses that will enable further studies of the relationships between cigarette smoking, the oral microbiome and tobacco-related cancers.

Under an Amendment, the participants will be contacted to provide another set of oral swabs and mouthwash samples. The goal is to examine the stability or oral microbiota in 3-6 months and confirm the results based on the first time point. The collection methods, assays and analyses will be analogous to those performed previously.

ELIGIBILITY:
* INCLUSION CRITERIA

This study will recruit a convenience sample of 50 volunteers (25 current smokers with at least 5 years of smoking history, 25 never smokers). Current smokers are defined as individuals who have smoked more than 100 cigarettes in their lifetime and have smoked 5 or more cigarettes in the last 24 hours. Recent use of other tobacco products (pipe, cigar, snuff, cigarillos, and chewing tobacco) is an overall exclusion, but use in the remote past (> 6 month ago) is acceptable in smokers. Never smokers are defined as individuals who have never smoked cigarettes nor used any other tobacco products including pipe, cigar, snuff, cigarillos, or chewing tobacco.

The ethnic mix of the clinic is roughly 50% Caucasians and 50% African- Americans with a small number of unspecified or other racial groups. The median age is about 50 and the gender mix consists of an equal number of men and women. We therefore will select smokers and frequency match to non-smokers based on ethnicity (White, African-American), gender (male, female), and age (above or below the median, estimated to be 50).

EXCLUSION CRITERIA

We will exclude pregnant women and other racial groups because they may represent very small numbers and thus be difficult to match. Hormonal changes associated with pregnancy and unique cultural habits associated with specific ethnic groups could be associated with highly unique or variable microbiome patterns, and therefore reduce the power to detect differences associated with smoking which is our primary goal. We will also exclude subjects with antibiotic usage in the last three months and subjects with previous diagnosed major periodontal disease or cancer because they might be potential confounders.

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adult volunteers who attended a dental clinic at University of Rochester NY
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2013-05-23 (Actual); Primary Completion 2014-12-05 (Actual); Study Completion 2020-06-26 (Actual)

PRIMARY OUTCOMES:
This is a pilot study to demonstrate the effects of smoking on oralmicrobiotas across differenct oral cavity sites | ongoing
  This was a descriptive study involving ~ 25 smokers and 25 non-smokers. We found and published in 2017 that alpha diversity was lower in smokers than in nonsmokers in the buccal mucosa, but inother sample sites, microbial diversity and compositionwere not significantly different by smoking status.

CONTACTS AND LOCATIONS:
Overall Officials: Neil E Caporaso, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- University of Rochester, Rochester, New York, United States

REFERENCES:
- [Background] Human Microbiome Project Consortium. Structure, function and diversity of the healthy human microbiome. Nature. 2012 Jun 13;486(7402):207-14. doi: 10.1038/nature11234. PMID 22699609
- [Background] Stampfli MR, Anderson GP. How cigarette smoke skews immune responses to promote infection, lung disease and cancer. Nat Rev Immunol. 2009 May;9(5):377-84. doi: 10.1038/nri2530. PMID 19330016
- [Background] Segata N, Haake SK, Mannon P, Lemon KP, Waldron L, Gevers D, Huttenhower C, Izard J. Composition of the adult digestive tract bacterial microbiome based on seven mouth surfaces, tonsils, throat and stool samples. Genome Biol. 2012 Jun 14;13(6):R42. doi: 10.1186/gb-2012-13-6-r42. PMID 22698087